CLINICAL TRIAL: NCT01622751
Title: Plasma Adiponectin Level and Sleep Structures in Children With Prader-Willi Syndrome
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Other Study IDs: 2006-09-055
Record Dates: First submitted 2012-01-18; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Prader-Willi Syndrome; Obesity
Keywords: REM sleep; Adiponectin; Prader-Willi syndrome
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Context: Adiponectin is an adipose tissue-derived hormone with an insulin sensitizing effect, and has been related to obstructive sleep apnea syndrome. In addition, children with Prader-Willi syndrome (PWS) suffer from excessive daytime sleepiness and the abnormality of rapid eye movement (REM) sleep.

Objective: To determine if the sleep stages are related to the plasma levels of adiponectin, resistin, and RBP4 (retinol binding protein-4), and whether these relationships are influenced by age, obesity and insulin resistance.

DETAILED DESCRIPTION:
This comparative study was carried out in 28 PWS children and 18 controls. The enrolled PWS children were volunteers out of a pool of approximately 100 PWS children followed at Samsung Medical Center [median age 8.0 years, interquartile range (7.0-10.5 years), BMI: median 24.2 kg/m2 (23.0-27.5 kg/m2)] and 18 obese healthy children [median age 9.0 years interquartile range (7.0-11.0 years), BMI: median 24.2 kg/m2 interquartile range (23.1-27.6 kg/m2)].

ELIGIBILITY:
Inclusion Criteria:

* Prader Willi syndrome healthy children

Exclusion Criteria:

* history of seizure,
* mental or brain illness,
* adenoidectomy,
* tonsillectomy,
* craniofacial anomalies and any treatment at the time of the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population comprised 28 children with PWS and 18 controls. The enrolled children with PWS were volunteers from a pool of approximately 100 children with PWS followed up at the Samsung Medical Center. The controls were healthy children from several elementary and middle schools located in the southern areas of Seoul.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2007-01; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Kyu Jin, M.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine